CLINICAL TRIAL: NCT03671408
Title: Levels of High-Sensitivity C-Reactive Protein in Heart Transplant Patients With and Without Periodontitis
Brief Title: Levels of High-Sensitivity C-Reactive Protein in Heart Transplant Patients
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yasemin Sezgin, asistant professor, Baskent University
Other Study IDs: BaskentU3
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Heart Transplant Failure; Periodontitis; Crp
Keywords: heart transplant; periodontitis; hsCRP
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- periodontitis: periodontitis patients which were diagnosed based on clinical parameters
  Interventions: Other: clinical measurements
- gingivitis/healthy: gingivitis healthy patients which were diagnosed based on clinical parameters
  Interventions: Other: clinical measurements

INTERVENTIONS:
Other: clinical measurements — only clinical parameters were recorded
  Other Names: no intervention was made

SUMMARY:
Objectives: The outcomes of heart transplantation are very favorable but inflammation still plays a critical role in deterioration of chronic transplants. Periodontal diseases are not only limited to supporting structures of the teeth, they also cause systemic inflammation. Based on the importance of inflammation in heart transplant recipients and the association between periodontal disease and systemic inflammation, this study explored whether periodontitis may be a modifier of serum high-sensitivity C-reactive protein (HsCRP) in heart transplant patients.

ELIGIBILITY:
Inclusion Criteria:

be clinically stable be at least 1 year post-transplant; no history of antibiotic use during the preceding 4 months have had no periodontal treatment within the previous year.

Exclusion Criteria:

having other systemic infections

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who underwent heart transplant between 2004 and April 2016 at Baskent University Hospital,will be asked to participate in the study during routine outpaient visits at Baskent University Hospital
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
hscrp levels | day 1
  serum hscrp levels were compared between the groups

IPD SHARING:
Plan to Share IPD: No